CLINICAL TRIAL: NCT00900146
Title: Dose Finding, Safety and Efficacy of Monthly Subcutaneous Canakinumab Administration for the Treatment of Hyperglycemia in Metformin Monotherapy Treated Type 2 Diabetic Patients: a Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study
Brief Title: Dose Finding, Safety and Efficacy of Monthly Subcutaneous Canakinumab Administration in Metformin Monotherapy Treated Type 2 Diabetic Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Numerically modest lowering of HbA1c with canakinumab in combination with metformin was inadequate to continue patients with T2DM into Period IV of this study.
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885I2202
Record Dates: First submitted 2009-05-06; First posted 2009-05-12 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; canakinumab
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — canakinumab; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Canakinumab 5 mg + Metformin (Experimental): In 4-Month Dose-finding period, patients visited the clinic monthly and had 5 mg Canakinumab injected in the clinic at each visit and continued on a stable dose of metformin ≥ 1000 mg daily (or lower dose if required by local regulations). During this period, patients with consecutive morning fasting glucose >200 mg/dL were treated with a daily injection of insulin glargine as add-on therapy.
  The intermediate period began after patients completed their 4-month visit and lasted until the primary analysis was completed and the optimal dose was selected. Patients continued on their randomized treatment and made brief visits to the clinic every month. From this point onward, patients with consecutive HbA1c >7.5% were treated with a daily injection of insulin glargine as add-on therapy.
  Interventions: Drug: Canakinumab; Drug: Metformin
- Canakinumab 15 mg + Metformin (Experimental): In 4-Month Dose-finding period, patients visited the clinic monthly and had 15 mg Canakinumab injected in the clinic at each visit and continued on a stable dose of metformin ≥ 1000 mg daily (or lower dose if required by local regulations). During this period, patients with consecutive morning fasting glucose >200 mg/dL were treated with a daily injection of insulin glargine as add-on therapy.
  The intermediate period began after patients completed their 4-month visit and lasted until the primary analysis was completed and the optimal dose was selected. Patients continued on their randomized treatment and made brief visits to the clinic every month. From this point onward, patients with consecutive HbA1c >7.5% were treated with a daily injection of insulin glargine as add-on therapy.
  Interventions: Drug: Canakinumab; Drug: Metformin
- Canakinumab 50 mg + Metformin (Experimental): In 4-Month Dose-finding period, patients visited the clinic monthly and had 50 mg Canakinumab injected in the clinic at each visit and continued on a stable dose of metformin ≥ 1000 mg daily (or lower dose if required by local regulations). During this period, patients with consecutive morning fasting glucose >200 mg/dL were treated with a daily injection of insulin glargine as add-on therapy.
  The intermediate period began after patients completed their 4-month visit and lasted until the primary analysis was completed and the optimal dose was selected. Patients continued on their randomized treatment and made brief visits to the clinic every month. From this point onward, patients with consecutive HbA1c >7.5% were treated with a daily injection of insulin glargine as add-on therapy.
  Interventions: Drug: Canakinumab; Drug: Metformin
- Canakinumab 150 mg + Metformin (Experimental): In 4-Month Dose-finding period, patients visited the clinic monthly and had 150 mg Canakinumab injected in the clinic at each visit and continued on a stable dose of metformin ≥ 1000 mg daily (or lower dose if required by local regulations). During this period, patients with consecutive morning fasting glucose >200 mg/dL were treated with a daily injection of insulin glargine as add-on therapy.
  The intermediate period began after patients completed their 4-month visit and lasted until the primary analysis was completed and the optimal dose was selected. Patients continued on their randomized treatment and made brief visits to the clinic every month. From this point onward, patients with consecutive HbA1c >7.5% were treated with a daily injection of insulin glargine as add-on therapy.
  Interventions: Drug: Canakinumab; Drug: Metformin
- Placebo + Metformin (Placebo Comparator): In 4 month dose finding period as well as during intermediate period, patients received one injection of canakinumab matching placebo monthly and continued on a stable dose of metformin ≥ 1000 mg daily (or lower dose if required by local regulations).
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — Canakinumab lyophilized cake (25 mg and 150 mg in individual 6 mL glass vials ) was reconstituted and then used to dilute the 25mg or 150mg solutions to make 5mg, 15mg and 50mg injections.
  Arms: Canakinumab 15 mg + Metformin; Canakinumab 150 mg + Metformin; Canakinumab 5 mg + Metformin; Canakinumab 50 mg + Metformin
Drug: Metformin — Before randomization, in drug naïve patients at a dose of 1000 mg with the evening meal or 500 mg b.i.d. (twice daily) with two main meals. At the randomization visit, patients were prescribed with no less than 1,000mg/day.
Drug: Placebo — Placebo lyophilized cake will be reconstituted and then used to dilute the 25mg or 150mg solutions to make 5mg, 15mg and 50mg injections.
  Arms: Placebo + Metformin

SUMMARY:
This was a four month dose ranging study followed by a 24 to 48 month extension at the selected dose to characterize the safety and efficacy of the injectable IL-1B (interleukin 1, beta) antagonist canakinumab in the treatment of patients with Type 2 diabetes mellitus (T2DM) already treated on maximum dose metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a documented diagnosis of Type 2 diabetes confirmed by World Health Organization (WHO) criteria either a FPG≥ 7.0 mmol/l (126 mg/dl) or an Oral glucose tolerance test (OGTT) test 2-hour PG ≥ 11.1 mmol/l (200 mg/dl).
2. Patients must:

   * be naïve to anti-diabetes drug therapy (except for short term treatment courses with insulin in connection with hospitalization, etc.)
   * meet protocol specified Glycosylated hemoglobin / hemoglobin A1c (HbA1c) criteria
   * be eligible for metformin monotherapy OR
   * be on stable metformin monotherapy treatment for at least three months at Screening
   * meet protocol specified HbA1c criteria
   * take metformin as their first and only treatment with anti-diabetes drug therapy OR
   * be taking an AGI as their first and only anti-diabetes drug therapy (except short term treatment courses with insulin in connection with hospitalizations, etc)
   * meet protocol specified HbA1c criteria
   * be eligible for metformin monotherapy
3. Patients must have a morning fasting plasma glucose result < 180 mg/dl at Visit 3 (Month -1) analyzed by the Central Laboratory.
4. Were on a daily dose of metformin ≥ 1000 mg (or less according to local regulations)

Exclusion Criteria:

1. Type 1 diabetes, diabetes resulting from pancreatic injury or secondary forms of diabetes.
2. Any of the following significant laboratory abnormalities:

   * Serum Glutamic acid decarboxylase (GAD)-antibody positivity
   * Clinically significant Thyroid stimulating hormone (TSH) outside of normal range at Screening
   * Renal function indicating high risk metformin use, including serum creatinine concentrations (≥1.5 mg/dL for males, ≥1.4 mg/dL for females) or other evidence of abnormal creatinine clearance.
   * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2 x upper limit of normal (ULN), or total bilirubin > 2 x ULN and/or direct bilirubin > ULN at Screening, confirmed with repeat measure within one week.
3. History or current findings of active pulmonary disease as evidenced by a history of positive purified protein derivative (PPD), QuantiFERON-TB Gold (QFT-G), AFB sputum or positive PPD followed by positive chest x-ray or QFT-G, or ongoing antibiotic treatment for latent TB.
4. Risk factors for TB as defined in protocol
5. Known presence or suspicion of active or recurrent bacterial, fungal or viral infection at the time of enrollment proven or suspected to be related to immunocompromise including HIV or active or recurrent Hepatitis B and Hepatitis C.
6. Systemic or local treatment of any immune modulating agent in doses with systemic effects or live vaccinations within 3 months
7. Stroke, myocardial infarction, acute coronary syndrome, revascularization procedure or recurrent TIA within the last 6 months.
8. Unwillingness to use insulin glargine as the additional medication should glycemic control deteriorate.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2009-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corporation, Study Director — Sponsor GmbH
Locations (104):
- United States (18):
  - Anasazi Internal Medicine, Phoenix, Arizona
  - Whittier Institute of Diabetes, La Jolla, California
  - Novartis Investigative Site, Los Gatos, California
  - Novartis Investigative Site, Santa Monica, California
  - Orange County Research Center, Tustin, California
  - Novartis Investigative Site, Atlanta, Georgia
  - Deaconess Clinic, Evansville, Indiana
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Trenton, New Jersey
  - Diabetes Research Center, Columbus, Ohio
  - Tri-State Medical Group, Beaver, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Columbia, South Carolina
  - R/D Clinical Research, Lake Jackson, Texas
  - Novartis Investigative Site, Pasadena, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Medical Research Initiatives Inc, Virginia Beach, Virginia
- Argentina (8):
  - DIM Clinica Privada, Buenos Aires, Buenos Aires
  - Centro Medico Viamonte, Buenos Aires, Buenos Aires
  - Consultorios Asociados de Endocrinologia, Buenos Aires, Buenos Aires
  - Clinica de Fracturas y Ortopedia, Mar del Plata, Buenos Aires
  - Hospital Juan Ramon Vidal, Corrientes, Corrientes Province
  - Instituto de Investigaciones Biomedicas, Santa Fe, Santa Fe Province
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, Rosario Santa Fe
- Belgium (3):
  - Private Practice - DEMEULEMEESTER, Gozée
  - Novartis Investigative Site, Heist-op-den-Berg
  - UZ Brussel, Jette
- Novartis Investigative Site, Hong Kong, China
- Germany (15):
  - Praxis F. Franzmann, Bad Oeynhausen
  - emovis GmbH, Berlin
  - Praxis Dr. Stütz, Bretten
  - GWT-TUB GmbH, Dresden
  - Gemeinschaftspraxis und Dialysezentrum Karlstraße, Düsseldorf
  - Asklepios Klinik St. Georg, Hamburg
  - Städt. Kankenhaus Nordstadt, Hanover
  - Diabeteszentrum Hohenmölsen, Hohenmölsen
  - Johannes Gutenberg-Universität Mainz, Mainz
  - Zentrum für Klinische Forschung Neuwied (ZKSN), Neuwied
  - Praxis Dr. Wunderer, Nuremberg
  - Praxis Dr. Kosch, Pirna
  - Praxis Dr. Alawi, Saarlouis
  - Praxis Dr. Klein, Schenklengsfeld
  - Forschungszentrum Ruhr, KliFoCenter GmbH, Witten
- Hungary (6):
  - Fővárosi Önkormányzat Péterfy Sándor Utcai Kórház - Rendelőintézet és Baleseti Központ, Budapest
  - Sandor Karolyi Hospital, Budapest
  - Semmelweiss Medical University, Budapest
  - Kenezy Gyula Korhaz, Debrecen
  - Szegedi Egyetem, Szeged
  - Zala Megyei Korhaz, Zalaegerszeg
- India (12):
  - Bangalore Diabetes Hospital, Bangalore
  - Gokula Metropolis Clinical Research Centre, Bangalore
  - Jnana Sanjeevini Medical Center, Bangalore
  - SAMATVAM, Bangalore
  - Madras Diabetes Reasearch Foundation, Chennai
  - Nizam's Institute of Medical Sciences, Hyderabaad
  - Diabetes Thyroid Hormone Research Institute Pvt. Ltd., Indore
  - S R Kalla Memorial Gastro & General Hospital, Jaipur
  - Amrita Institute of Medical Sciences and Research Center, Kochi
  - Pitale Diabetes & Hormone Centre, Nagpur
  - Health and Research Centre, Trivandrum
  - King George Hospital, Visakhapatnam
- Japan (12):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - Kyushu Rosai Hospital, Kitakyushu, Fukuoka
  - NHO Yokohama Medical Center, Yokohama, Kanagawa
  - Musashikoganei Clinic, Koganei, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Fujikoshi Hospital, Toyama, Toyama
  - Kokura Medical Center, Kitakyushu
  - Seino Internal Medicine Clinic, Kōriyama
  - Geriatrics Research Institute Hospital, Maebashi
  - Takagi Hospital, Ohkawa
  - Sakai Hospital Kinki University School of Medicine, Sakai
- Peru (4):
  - Instituto Delgado de Investigacion Medica, Arequipa
  - Clinica Chiclayo, Chiclayo
  - Hospital Nacional Cayetano Heredia, San Martín de Porres
  - Centro de Investigacion Clinica Trujillo, Trujillo
- Romania (4):
  - Ambulatory of Institute of Nutrition Diseases and Diabetes, Bucharest
  - Medical Centre "Sanatatea ta", Bucharest
  - Novartis Investigative Site, Bucharest
  - Policlinica Dr. Citu Timisoara, Timișoara
- South Africa (7):
  - 203 Maxwell Centre, Durban
  - Parklands Medical Centre, Durban
  - St Augustines Medical Centre, Durban
  - Synapta Clinical Research Centre, Durban
  - Drs Essack and Mitha, Johannesburg
  - 26 Daffodil Street, KwaDukuza
  - PE Greenacres Hospital, Port Elizabeth
- South Korea (3):
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Suwon
- Turkey (Türkiye) (7):
  - Ankara Ataturk Training and Research Hospital, Ankara
  - Gulhane Askeri Tip Akademisi, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - S.B. Yildirim Beyazit Training and Research Hospital, Ankara
  - Istanbul University Cardiology Institute, Istanbul
  - Ege University Medical Faculty, Izmir
  - Hayat Tip Merkezi (Hayat Medical Center) Deapartment of Internal Diseases, Karabük
- United Kingdom (4):
  - Morriston Hospital, Swansea, England
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Rowden Medical Partnership, Wiltshire

REFERENCES:
- [Derived] Noe A, Howard C, Thuren T, Taylor A, Skerjanec A. Pharmacokinetic and pharmacodynamic characteristics of single-dose Canakinumab in patients with type 2 diabetes mellitus. Clin Ther. 2014 Nov 1;36(11):1625-37. doi: 10.1016/j.clinthera.2014.08.004. Epub 2014 Sep 18. PMID 25240532
- [Derived] Hensen J, Howard CP, Walter V, Thuren T. Impact of interleukin-1beta antibody (canakinumab) on glycaemic indicators in patients with type 2 diabetes mellitus: results of secondary endpoints from a randomized, placebo-controlled trial. Diabetes Metab. 2013 Dec;39(6):524-31. doi: 10.1016/j.diabet.2013.07.003. Epub 2013 Sep 25. PMID 24075453
- [Derived] Ridker PM, Howard CP, Walter V, Everett B, Libby P, Hensen J, Thuren T; CANTOS Pilot Investigative Group. Effects of interleukin-1beta inhibition with canakinumab on hemoglobin A1c, lipids, C-reactive protein, interleukin-6, and fibrinogen: a phase IIb randomized, placebo-controlled trial. Circulation. 2012 Dec 4;126(23):2739-48. doi: 10.1161/CIRCULATIONAHA.112.122556. Epub 2012 Nov 5. PMID 23129601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study consisted of four periods: screening (Period I), dose-finding (Period II), intermediate (Period III),and long-term continuation (Period IV). Eligible patients were randomized for 4-month treatment of Period II. Intermediate period continued until primary analysis was completed and optimal dose was selected. Study got terminated in Period III.
Pre-assignment Details: A total of 556 patients were randomized in Period II. 5 patients one in each 5, 15, 50mg Canakinumab arms and 2 in Placebo were randomized in error, but never received study treatment. All tables reflect the 551 treated patients.
Period: Dose Finding: Period II (4 Months)
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Started | 93 | 95 | 92 | 92 | 179
Full Analysis Set (FAS)/Safety | 93 | 95 | 92 | 92 | 179
Completed | 88 | 93 | 87 | 90 | 167 (Placebo also included 1 patient with no study completion page.)
Not Completed | 5 | 2 | 5 | 2 | 12
Not completed — Withdrawal by Subject | 2 | 2 | 5 | 1 | 9
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 3
Not completed — Administrative problems | 1 | 0 | 0 | 0 | 0
Period: Intermediate: Period III
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Started | 87 | 93 | 84 | 90 | 167
Safety Set | 86 | 92 | 84 | 90 | 166
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 87 | 93 | 84 | 90 | 167
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 3
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 1
Not completed — Administrative problems | 85 | 92 | 84 | 90 | 163

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin | Total
Number analyzed (Participants) | 93 | 95 | 92 | 92 | 179 | 551
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measures were based on the full analysis set (FAS) which included all randomized patients except for mis-randomized patients. Mis-randomized patients referred to patients who are not qualified for randomization but who were inadvertently randomized into the study and did not receive study drug.
  years | 53.5 (10.27) | 55.5 (9.70) | 53.0 (9.29) | 53.7 (10.36) | 54.3 (10.15) | 54.1 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 46 | 47 | 35 | 74 | 240
  Male | 55 | 49 | 45 | 57 | 105 | 311

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events, Death and Clinical Significant AEs During 4 Months (Period II)
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: 4 months (Period II)
Population: The safety set (SAF) included all patients who received at least one dose of study medication during Period II.
Measure: Number; unit: Participants
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 93 | 95 | 92 | 92 | 179
Participants
  Any Adverse Events | 33 | 43 | 45 | 43 | 76
  Death | 0 | 0 | 0 | 0 | 0
  Serious Adverse Events | 2 | 1 | 2 | 5 | 6

2. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Month 4 During Dose-finding Period of the Study (Period II)
Description: HbA1c was measured by National glycohemoglobin standardization program (NGSP) certified methodology. HbA1c is an integrated measure of average glucose concentration in plasma in the last 2-3 months. The analysis of covariance (ANCOVA) included treatment and metformin dose group as main effects and baseline HbA1c as a covariate.
Time Frame: Baseline, Month 4
Population: The full analysis set (included all randomized patients except for mis-randomized patients who randomized in error but did not receive study drug. Last observation carried forward (LOCF) method was used for patients without Month 4 HbA1c data for any reason and who used rescue medication or any other glucose lowering agents other than metformin.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin A1c
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 92 | 94 | 89 | 91 | 175
percentage of hemoglobin A1c | -0.19 (0.072) | -0.29 (0.071) | -0.31 (0.073) | -0.25 (0.071) | -0.13 (0.053)

3. Secondary Outcome: Change From Baseline in C-peptide Area Under Curve (AUC 0-4 Hours ) Following Meal Test (Period II)
Description: A standard liquid mixed-meal challenge was done at baseline and Month 4. Patients completed each standard meal challenge with measurement of C-peptide prior to and after a liquid mixed meal. Sampling times were -20, -10, and -1, 10, 20, 30, 60, 90, 120, 150, 180 and 240 minutes relative to start of meal. C-peptide levels over 4 hrs were shown as Area Under the Curve,(AUC). AUC was calculated as: x=1 AUC ΣAx n Where Ax = AUC for the 240 min.interval, and X = 1 for the 1st interval. The analysis of covariance included baseline C-peptide AUC 0-4 hours as a covariate.
Time Frame: Baseline, Month 4
Population: The full analysis set included all randomized patients except for mis-randomized patients who inadvertently randomized into study and did not receive study drug. Last observation carried forward method was used for patients without Month 4 data for any reason and who used rescue medication or any other glucose lowering agents other than metformin.
Measure: Least Squares Mean (Standard Error); unit: nmol*hour/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 81 | 87 | 83 | 91 | 153
nmol*hour/L | -0.399 (0.1444) | -0.388 (0.1394) | -0.834 (0.1425) | -0.610 (0.1396) | -0.588 (0.1070)

4. Secondary Outcome: Change From Baseline in Prandial Plasma Glucose Area Under Curve (AUC0-4 Hours ) Following Meal Test (Period II)
Description: A standard liquid mixed-meal challenge was done at baseline and Month 4. Patients completed each standard meal challenge with measurement of glucose prior to and after a liquid mixed meal. Sampling times were -20, -10, and -1, 10, 20, 30, 60, 90, 120, 150, 180 and 240 minutes relative to the start of meal. Glucose levels over 4 hrs were shown as Area Under the Curve,(AUC). AUC was calculated as: x=1 AUC ΣAx n Where Ax = AUC for the 240 min.interval, and X = 1 for the 1st interval. The model of analysis of covariance included baseline plasma glucose AUC 0-4 hours as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol*hour/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 79 | 83 | 82 | 84 | 147
mmol*hour/L | -0.999 (0.8094) | -1.012 (0.7917) | -2.103 (0.7928) | 1.618 (0.7791) | -0.851 (0.6053)

5. Secondary Outcome: Change From Baseline in Insulin Area Under Curve (AUC 0-4 Hours ) Following Meal Test (Period II)
Description: A standard liquid mixed-meal challenge was done at baseline and Month 4. Patients completed each standard meal challenge with measurement of insulin prior to and after a liquid mixed meal. Sampling times were -20, -10, and -1, 10, 20, 30, 60, 90, 120, 150, 180 and 240 minutes relative to the start of meal. Insulin levels over 4 hrs were shown as Area Under the Curve,(AUC). AUC was calculated as: x=1 AUC ΣAx n Where Ax = AUC for the 240 min.interval, and X = 1 for the 1st interval. Model of analysis of covariance included baseline insulin AUC 0-4 hours as covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol*hour/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 68 | 73 | 70 | 77 | 133
pmol*hour/L | 18.623 (28.5445) | 66.237 (27.4053) | -14.016 (27.9738) | -20.583 (26.5602) | 0.121 (20.7195)

6. Secondary Outcome: Change From Baseline in 2-hour Glucose Level Following Meal Test (Period II)
Description: A standard liquid mixed-meal challenge was done at baseline and Month 4. Patients fasted overnight after 10 pm on day prior to scheduled visit. Study visits should occur before 10 am. Patients completed each standard meal challenge with measurement of glucose prior to and after a liquid mixed meal. The sampling times were -20, -10, and -1, 10, 20, 30, 60, 90, 120, 150, 180 and 240 minutes relative to the start of meal. The analysis of covariance included treatment and metformin dose group as main effects and baseline 2-hour glucose level as covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 79 | 85 | 83 | 84 | 151
mmol/L | -0.427 (0.2537) | -0.239 (0.2457) | -0.777 (0.2471) | 0.262 (0.2445) | -0.347 (0.1873)

7. Secondary Outcome: Change From Baseline in Peak Glucose Level Following Meal Test (Period II)
Description: A standard liquid mixed-meal challenge was done at baseline and Month 4. Patients fasted overnight after 10 pm on day prior to scheduled visit. Study visits should occur before 10 am. Patients completed each standard meal challenge with measurement of glucose prior to and after a liquid mixed meal. The sampling times were -20, -10, and -1, 10, 20, 30, 60, 90, 120, 150, 180 and 240 minutes relative to the start of meal. The analysis of covariance included treatment and metformin dose group as main effects and baseline peak glucose level as covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 81 | 85 | 83 | 87 | 152
mmol/L | -0.386 (0.2302) | -0.380 (0.2257) | -0.565 (0.2270) | 0.381 (0.2208) | -0.339 (0.1711)

8. Secondary Outcome: Change From Baseline in Peak C-peptide Following Meal Test (Period II)
Description: A standard liquid mixed-meal challenge was done at baseline and Month 4. Patients fasted overnight after 10 pm on the day prior to scheduled visit. Study visits should occur before 10 am. Patients completed each standard meal challenge with measurement of C-peptide prior to and after a liquid mixed meal. Sampling times were -20, -10, and -1, 10, 20, 30, 60, 90, 120, 150, 180 and 240 minutes relative to the start of meal. The analysis of covariance included treatment and metformin dose group as main effects and baseline peak C-peptide level as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 84 | 89 | 84 | 89 | 154
nmol/L | -0.075 (0.0524) | -0.115 (0.0509) | -0.227 (0.0523) | -0.207 (0.0506) | -0.212 (0.0394)

9. Secondary Outcome: Change From Baseline in Peak Insulin Level Following Meal Test (Period II)
Description: A standard liquid mixed-meal challenge was done at baseline and Month 4. Patients fasted overnight after 10 pm on day prior to scheduled visit. Study visits should occur before 10 am. Patients completed each standard meal challenge with measurement of insulin prior to and after a liquid mixed meal. The sampling times were -20, -10, and -1, 10, 20, 30, 60, 90, 120, 150, 180 and 240 minutes relative to the start of meal. The analysis of covariance included treatment and metformin dose group as main effects and baseline 2-hour insulin level as covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 76 | 81 | 82 | 84 | 148
pmol/L | 13.1 (14.40) | 26.0 (14.00) | 2.0 (13.88) | -7.0 (13.61) | 1.7 (10.59)

10. Secondary Outcome: Change From Baseline in Insulin Secretion Rates Relative to Glucose AUC (0-2 Hours) at Month 4 Following Meal Test (Period II)
Description: Change in Insulin Secretion Rate stimulated by Liquid mixed-meal challenge. A standard liquid mixed-meal challenge was done at baseline and Month 4. Blood samples were taken prior to and after meal for glucose and insulin at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes relative to the start of the meal. The model of analysis of covariance included baseline Insulin secretion rate relative to glucose AUC at 0-2 hours as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m²/mmol *hour/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 77 | 83 | 81 | 82 | 149
pmol/min/m²/mmol *hour/L | -0.369 (0.6922) | -0.331 (0.6705) | -1.761 (0.6744) | -2.428 (0.6681) | -1.635 (0.5084)

11. Secondary Outcome: Change From Baseline in 2 Hour Insulin Secretion Rate Derived Based on Glucose and C-peptide Following at Month 4 Following Meal Test (Period II)
Description: A standard liquid mixed-meal challenge was done at baseline and Month 4. A 2 hour insulin secretion rate using deconvolution was performed. The deconvolution was an algorithm that analyzed the insulin secretion rate relative to glucose and C-peptide combined. Blood samples were taken prior to and after meal at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes relative to the start of the meal. The analysis of covariance included treatment and metformin dose group as main effects and baseline 2 hour Insulin secretion rate as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m²
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 80 | 88 | 83 | 86 | 152
pmol/min/m² | -17.022 (10.4317) | -9.607 (9.9815) | -31.296 (10.2302) | -38.515 (10.0176) | -24.812 (7.6980)

12. Secondary Outcome: Change From Baseline in Peak Plasma Glucose Level (7-point Glucose Testing) at Month 4(Period II)
Description: Patients were asked to check their glucose level (7 times) using their glucose meter on one of the seven days prior to the Meal Challenge Visits (Period II: baseline, Month 4. Patient was instructed to test at following timepoints: fasting before breakfast, 2 hours after starting breakfast, before lunch, 2 hours after starting lunch, before dinner, 2 hours after dinner and at bedtime. The patient documented the results in their Study Diary. The analysis of covariance included treatment and metformin dose group as main effects and baseline peak plasma glucose level as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 81 | 85 | 82 | 86 | 152
mmol/L | -0.549 (0.2669) | -0.129 (0.2610) | -0.421 (0.2653) | -0.333 (0.2578) | -0.212 (0.1975)

13. Secondary Outcome: Change From Baseline in Average Plasma Glucose Level (7-point Glucose Testing) at Month 4 (Period II)
Description: Patients were asked to check their glucose level (7 times) using their glucose meter on one of the seven days prior to the Meal Challenge Visits (Period II: Month 0 (Baseline), Month 4. Patient was instructed to test at following timepoints: fasting before breakfast, 2 hours after starting breakfast, before lunch, 2 hours after starting lunch, before dinner, 2 hours after dinner and at bedtime. Patient documented the results in their Study Diary. The analysis of covariance included treatment and metformin dose group as main effects and baseline average plasma glucose level as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 81 | 85 | 82 | 86 | 152
mmol/L | -0.357 (0.1626) | -0.218 (0.1589) | -0.275 (0.1614) | -0.040 (0.1569) | -0.091 (0.1203)

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Month 4 (Period II)
Description: Change in Fasting Glucose Level measured from plasma taken at Baseline and at Month 4. The analysis of covariance included treatment and metformin dose group as main effects and baseline fasting plasma glucose level as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 89 | 93 | 88 | 90 | 172
mmol/L | 0.25 (0.162) | -0.19 (0.159) | -0.29 (0.162) | 0.19 (0.160) | 0.01 (0.118)

15. Secondary Outcome: Change From Baseline in Fasting Insulin at Month 4 (Period II)
Description: Change in fasting insulin Level measured from blood samples taken at Baseline and at Month 4. The analysis of covariance included treatment and metformin dose group as main effects and baseline fasting insulin level as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 75 | 81 | 77 | 83 | 143
pmol/L | 4.3 (4.74) | 7.2 (4.57) | 7.0 (4.67) | 4.4 (4.47) | -0.4 (3.50)

16. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment B (HOMA2 B) Beta Cell Function (%B) at Month 4 (Period II)
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance and beta (β)-cell function. HOMA2-B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state beta cell function (%B) as a percentage of a normal reference population (normal young adults). Time profile of postprandial glucose, insulin and C-peptide were assessed as measures of β-cell response to stimulation. The analysis of covariance included treatment and metformin dose group as main effects and baseline HOMA-B as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of beta cell function
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 75 | 79 | 77 | 83 | 143
percentage of beta cell function | -1.067 (6.0549) | 2.259 (5.9304) | 8.215 (5.9727) | 6.217 (5.7307) | -2.182 (4.4846)

17. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment Insulin Resistance (HOMA2 IR) at Month 4 (Period II)
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance and beta (β)-cell function. HOMA2-IR is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin resistance which is the reciprocal of insulin sensitivity (%S)(100/%S)as a percentage of a normal reference population (normal young adults). The analysis of covariance included treatment and metformin dose group as main effects and baseline HOMA2 IR as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of insulin resistance
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 75 | 81 | 77 | 83 | 143
percentage of insulin resistance | 0.245 (0.3107) | 0.517 (0.2990) | 0.255 (0.3054) | 0.252 (0.2925) | 0.013 (0.2286)

18. Secondary Outcome: Change From Baseline in Quantitative Insulin Sensitivity Check Index (QUICKI) at Month 4 (Period II)
Description: The Quantitative Insulin Sensitivity Check Index (QUICKI) score, measures insulin sensitivity which is the inverse of insulin resistance. The score is calculated by the equation: 1 /(log(fasting insulin µU/mL) + log(fasting glucose mg/dL)). In normal subjects, the mean score ± SE is 0.366 ± 0.029. The analysis of covariance included treatment and metformin dose group as main effects and baseline QUICKI as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 75 | 81 | 77 | 83 | 143
units on a scale | -0.001 (0.0017) | 0.000 (0.0016) | -0.003 (0.0017) | -0.001 (0.0016) | 0.000 (0.0013)

19. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP) at Month 4 (Period II)
Description: The change from baseline in hsCRP (on the logarithmic scale) at Month 4 was measured for this analysis. The analysis of covariance included treatment and metformin dose group as main effects and baseline hsCRP as a covariate.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: log (mg/L)
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 89 | 93 | 87 | 91 | 168
log (mg/L) | -0.19 (0.037) | -0.32 (0.036) | -0.44 (0.037) | -0.40 (0.036) | -0.08 (0.027)

20. Secondary Outcome: Percentage Change From Baseline in Fasting Lipids Profile at Month 4 (Period II)
Description: The fasting lipid profiles included triglycerides, total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), calculated very low-density lipoprotein (VLDL), non-HDL cholesterol. Percentage change was measured as [(value at month 4 - baseline value)/baseline value]*100%. The analysis of covariance model included treatment and metformin dose group as main effects and baseline triglycerides, total cholesterol, LDL, HDL, VLDL and non-HDL as covariates.
Time Frame: Baseline, Month 4
Population: The full analysis set included all randomized patients except for mis-randomized patients who randomized in error, did not receive study drug. LOCF method was used for patients without Month 4 data for any reason and who used rescue drug or any other glucose lowering agents other than metformin. 'n' = patients with baseline and endpoints data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 93 | 95 | 92 | 92 | 179
percent change
  Total cholesterol (n = 91, 93, 88, 91, 172) | 3.163 (1.5364) | 3.922 (1.5188) | 5.334 (1.5542) | 6.265 (1.5234) | 2.697 (1.1334)
  Triglycerides (n = 91, 93, 88, 91, 172) | 16.127 (4.3130) | 7.903 (4.2688) | 19.937 (4.3684) | 18.795 (4.2786) | 7.009 (3.1813)
  LDL (n = 90, 90, 85, 87, 165) | 2.624 (2.4606) | 4.741 (2.4582) | 2.705 (2.5137) | 5.938 (2.4752) | 5.129 (1.8351)
  HDL (n = 91, 93, 88, 91, 172) | 1.438 (1.6619) | 5.346 (1.6441) | 8.074 (1.6853) | 6.780 (1.6494) | 3.963 (1.2303)
  VLDL (n= 90, 90, 85, 87, 165) | 15.646 (3.9196) | 6.711 (3.9118) | 16.533 (3.9986) | 16.618 (3.9373) | 7.370 (2.9203)
  Non-HDL (n = 91, 93, 88, 91, 172) | 4.25 (2.022) | 4.40 (1.999) | 5.17 (2.046) | 7.25 (2.005) | 3.04 (1.491)

21. Primary Outcome: Change From Baseline in Dynamic Phase Secreted Insulin Per Unit of Glucose Concentration (Φd) Over 4 Months (Period III)
Description: This was planned as interim analysis and was not conducted because the study was terminated in period III.
Time Frame: Baseline, Over Month 4
Population: The benefit of canakinumab for the treatment of patients with type 2 diabetes mellitus in combination with metformin was inadequate to continue patients into Period IV in the present study, and therefore decided to terminate the study during Period III.
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m2/mmol* hour/L
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients have been exposed up to 15 months (median exposure however was at about 6 months)
Description: The data reported below in the safety tables are from the pooled Phase II and Phase III data.
Groups:
- Canakinumab 150 mg + Metformin: Experimental: Canakinumab 150 mg + Metformin In 4-Month Dose-finding period, patients visited the clinic monthly and had 150 mg Canakinumab injected in the clinic at each visit and continued on a stable dose of metformin ≥ 1000 mg daily (or lower dose if required by local regulations). During this period, patients with consecutive morning fasting glucose >200 mg/dL were treated with a daily injection of insulin glargine as add-on therapy.
  The intermediate period began after patients completed their 4-month visit and lasted until the primary analysis was completed and the optimal dose was selected. Patients continued on their randomized treatment and made brief visits to the clinic every month. From this point onward, patients with consecutive HbA1c >7.5% were treated with a daily injection of insulin glargine as add-on therapy.
Arm/Group | Canakinumab 5 mg + Metformin | Canakinumab 15 mg + Metformin | Canakinumab 50 mg + Metformin | Canakinumab 150 mg + Metformin | Placebo + Metformin
Serious Adverse Events (participants affected / at risk) | 3/93 | 1/95 | 5/92 | 7/92 | 8/179
Other Adverse Events (participants affected / at risk) | 9/93 | 9/95 | 15/92 | 8/92 | 26/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 5 mg + Metformin (N=93) | Canakinumab 15 mg + Metformin (N=95) | Canakinumab 50 mg + Metformin (N=92) | Canakinumab 150 mg + Metformin (N=92) | Placebo + Metformin (N=179)
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Graft infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 5 mg + Metformin (N=93) | Canakinumab 15 mg + Metformin (N=95) | Canakinumab 50 mg + Metformin (N=92) | Canakinumab 150 mg + Metformin (N=92) | Placebo + Metformin (N=179)
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 5 | 0 | 3
Nasopharyngitis (Infections and infestations) | 5 | 4 | 9 | 4 | 15
Urinary tract infection (Infections and infestations) | 3 | 4 | 5 | 5 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.